CLINICAL TRIAL: NCT05877378
Title: Efficacy of Single-use Negative Pressure Therapy With PICO System in Chronic Ulcers
Brief Title: Efficacy of PICO Single-use System in Chronic Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMCU001
Record Dates: First submitted 2023-05-11; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-01

CONDITIONS: Chronic Ulcer; Venous Ulcer; Diabetic Foot Ulcer; Pressure Injury
Keywords: negative pressure therapy; chronic wound; ulcer; conventional treatment
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot; Pressure Ulcer; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group measurements will be carried out every 7 days, since the PICO system lasts from 7 to 14 days, except when the ulcer presents infection, which will be cured every 2-3 days.
  Interventions: Device: Single-use negative pressure therapy (PICO)
- Control (No Intervention): The control group measurements will be carried out every 7 days, except when the ulcer is infected, when the cure will be carried out every 2-3 days. This group (GC) will be treated mainly with betadine and sugar, or other treatments such as alginate patches, corticosteroids, Aquacel, Celestoderm or Mepitel.

INTERVENTIONS:
Device: Single-use negative pressure therapy (PICO) — PICO system will be applied to patients in the intervention group with diabetic foot ulcers, venous leg ulcers or pressure ulcers. This device will be changed every 7 days, until the wound is closed, or until a set period of study duration, approximately 12 weeks.
  Arms: Intervention

SUMMARY:
A clinical trial will be carried out comparing the efficacy of PICO system based on negative pressure therapy (NPT) in adults with chronic ulcers compared to conventional treatments.

DETAILED DESCRIPTION:
Due to the current scientific and clinical evidence shows that NPT offers guarantees as complementary care, improving healing and reducing amputations in patients with chronic ulcers, treatment with PICO single-use NPT, should be considered as the first option.

This clinical trial include adults from the Hospital General Universitario of Toledo with 2 arms (intervention and control) and the intervention will last 12 weeks.

The intervention proposed in the study will consist of evaluating the decrease in size, the healing rate, the adverse effects and the quality of life related to the health of the patients compared with traditional treatments.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes over 18 years.
* Patients with chronic ulcers: venous leg ulcer, diabetic foot ulcer or pressure ulcers.
* Patients capable of complying with the protocol instructions and signing the informed consent (IC) or with limited capacity to act, in which case their relatives would be informed, who would be the ones who would grant the signed informed consent.
* Acceptable state of health.

Exclusion Criteria:

* Malignant ulcers.
* Ulcers with abundant exudate.
* Non-modifiable anatomical location to create hermetic seal of the dressing.
* Suspected or known allergy to components of TPN systems.
* Pregnancy.
* Serious cardiovascular diseases.
* Diagnosis of vasculitis or claudication.
* Current administration of systemic chemotherapy or corticosteroids.
* Having received prior treatment with TPN or hyperbaric oxygen in the 7 days prior to screening.
* Leukopenia, thrombocytopenia, anemia, increased bilirubin or three times the level of liver enzymes.
* Deep venous thrombosis.
* Refusal or inability to tolerate compression therapy, exposure of muscles, tendons or bone.
* Diagnosis of active Charcot foot syndrome.
* Malnutrition or eating disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in the size of wounds | 12 weeks
  The size of the wound will be measured by a nurse using a ruler every day that the patient goes to the cure to compare de first measure from the last one.
Healing time | 12 weeks
  The healing time will be measured by a nurse during the days of the treatment
Cure rate | 12 weeks
  The cure rate will be measured by a nurse during the days of the treatment
Number of participants with adverse effects | 12 weeks
  The nurse will observe how many patients may have adverse effects.
Health-related effects on quality of life. | 12 weeks
  Patients will answer the European Quality of Life-5 Dimension. This consists of a questionnaire to measure health-related quality of life, before and after the treatment. This scale have two parts: in the first one, 0 is the best score; and 15 is the worst. In the second part (that is a pain rating scale): 0 is the worst state of health imaginable and 10 the best state of health imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Celia Villalba Aguilar, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No